CLINICAL TRIAL: NCT04335357
Title: A One Year, Randomized, Double-Blind, Placebo-Controlled Study of TBR-760 in Adult Patients With Non-Functioning Pituitary Adenomas
Brief Title: TBR-760 in Adult Patients With Non-Functioning Pituitary Adenomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tiburio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBR-760-NFPA-201
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Non-Functional Pituitary Adenoma; Pituitary Tumor, Nonfunctioning
MeSH Terms: conditions — Pituitary Neoplasms | interventions — TBR-760

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The appearance and fill of placebo syringes will be identical to the active comparator.
  Interventions: Drug: Placebo
- TBR-760 (Active Comparator): TBR-760 is supplied as a ready-to-use solution in pre-filled syringes at a concentration of 5 mg/ml.
  Interventions: Drug: TBR-760

INTERVENTIONS:
Drug: TBR-760 — TBR-760 is intended for SC administration. The target dose to be studied in this study is 6 mg SC given once weekly.
  Arms: TBR-760
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, efficacy, PK, and PD of the chimeric dopamine-somatostatin receptor agonist, TBR-760, in adult patients with NFPA over 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, efficacy, PK, and PD of the chimeric dopamine-somatostatin receptor agonist, TBR-760, in adult patients with NFPA over 52 weeks. Approximately 150 patients will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of NFPA (defined as lack of clinical and biochemical evidence of adenohypophyseal hormone excess), and be status-post one TSS with a NFPA remnant of ≥ 10mm (maximum diameter)
* Study subjects must be capable of giving informed consent and reading and signing the informed consent form after the nature of the study has been fully explained by the Investigator or Investigator designee
* Study subject must be willing and able to complete all study assessments and procedures and to communicate effectively with the Investigator and site staff.

Key Exclusion Criteria:

* Has undergone more than one TSS, or had TSS <6 months prior to screening, or is anticipated to require TSS within 6 months of Screening
* Has undergone radiation therapy to the head for any reason, or is already planned to have or anticipated to require radiation therapy during the study period;
* Has any contraindications to magnetic resonance imaging including allergy or intolerance to gadolinium or gadolinium-based contrast;
* In the opinion of the Investigator, the patient is unable to meet the requirements of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
tumor volume reduction | 52 weeks
  the primary efficacy endpoint is the percentage of patients with tumor volume reduction

IPD SHARING:
Plan to Share IPD: No